CLINICAL TRIAL: NCT07213986
Title: Pilot Trial of the Vibrant Capsule for Spinal Cord Injury Neurogenic Bowel Dysfunction
Brief Title: Vibrant Capsule for Spinal Cord Injury Neurogenic Bowel Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mission Connect (Unknown)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-25-0364; Project# 0019646 (Other Grant/Funding Number: Misssion Connect)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Bowel Dysfunction; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vibrant Capsule (Experimental)
  Interventions: Device: Vibrant Capsule

INTERVENTIONS:
Device: Vibrant Capsule — The Vibrant capsule is designed to alleviate chronic constipation by stimulating the colon through gentle vibrations. The Vibrant capsule will be swallowed and tracked through the digestive system of spinal cord injury patients.

SUMMARY:
The goal of this study is to test the safety and effectiveness of Vibrant capsules in spinal cord injury patients with neurogenic bowel.

DETAILED DESCRIPTION:
The purpose of this study is to see how well the Vibrant capsule works at treating people with spinal cord injury (SCI)-induced upper motor neuron (UMN) neurogenic bowel. This study will test the safety of the Vibrant capsule. This Vibrant capsule has been approved by the Food and Drug Administration (FDA) for chronic idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic spinal cord injury (SCI) of more than one year.
* Stable neurological level and function of SCI for at least six months.
* Consistent bowel program without changes for at least 3 months.
* At least one scheduled bowel movement (BM) every three days.
* Use of digital stimulation, suppositories, enemas, or mini enemas, as part of the scheduled bowel program.
* Use of oral medications as part of the bowel program.

Exclusion Criteria:

* Bowel incontinence occurring more than once per week.
* Non-English-speaking individuals.
* History of bowel obstruction, ileus, diverticulitis, or bowel surgery for a disease (appendix removal is ok).
* Persistent autonomic dysreflexia (AD) triggered by bowel movements.
* Recent changes to spasticity medications within the past month.
* History of significant gastrointestinal disorders
* History of Zenker's diverticulum
* Dysphagia
* Esophageal stricture
* Eosinophilic esophagitis or achalasia
* Pregnancy.
* Presence of implanted devices that could be affected by proximity to a direct current magnetic field.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Vibrant capsule as indicated by number of participants who had an adverse event | baseline week 1, baseline week 2, baseline week 3, baseline week 4
Safety of Vibrant capsule as indicated by number of participants who had an adverse event | week 1 with treatment, week 2 with treatment, week 3 with treatment, week 4 with treatment
Safety of Vibrant capsule as assessed by the Penn Spasm Frequency Scale (PSFS) | baseline week 1, baseline week 2, baseline week 3, baseline week 4
  The total score on the Penn Spasm Frequency Scale (PSFS) ranges from 0 to 7, and a higher score indicates greater spasm frequency and severity.
Safety of Vibrant capsule as assessed by the Penn Spasm Frequency Scale (PSFS) | week 1 with treatment, week 2 with treatment, week 3 with treatment, week 4 with treatment
  The total score on the Penn Spasm Frequency Scale (PSFS) ranges from 0 to 7, and a higher score indicates greater spasm frequency and severity.
Safety as assessed by average weekly Numerical Pain Score | baseline week 1, baseline week 2, baseline week 3, baseline week 4
  The Numerical Pain Score ranges from 0 to 10, with a higher score indicating greater pain.
Safety as assessed by average weekly Numerical Pain Score | week 1 with treatment, week 2 with treatment, week 3 with treatment, week 4 with treatment
  The Numerical Pain Score ranges from 0 to 10, with a higher score indicating greater pain.
Safety as assessed by the Neurogenic Bladder Symptom Score (NBSS) | baseline, week 3
  The Neurogenic Bladder Symptom Score (NBSS) ranges from 0 to 96, with a higher score indicating greater Neurogenic Bladder Symptoms.
Safety as assessed by the Neurogenic Bladder Symptom Score (NBSS) | week 1 with treatment, week 4 with treatment
  The Neurogenic Bladder Symptom Score (NBSS) ranges from 0 to 96, with a higher score indicating greater Neurogenic Bladder Symptoms.

SECONDARY OUTCOMES:
Feasibility as indicated by the number of participants that adhere to the prescribed use of Vibrant | from week 1 with treatment to week 4 with treatment
  Feasibility of the Vibrant capsule will be recorded in this patient population by adherence to the protocol.
Feasibility of using the Vibrant capsule as indicated by a satisfaction survey | end of study (4 weeks after start of treatment)
  Feasibility will also be recorded by a satisfaction survey completed by the study participant. Total score ranges from 0 to 40, with a higher score indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Gastroenterology Chronic Constipation Task Force. An evidence-based approach to the management of chronic constipation in North America. Am J Gastroenterol. 2005;100 Suppl 1:S1-4. doi: 10.1111/j.1572-0241.2005.50613_1.x. No abstract available. PMID 16008640
- [Background] Rao SSC, Lembo A, Chey WD, Friedenberg K, Quigley EMM. Effects of the vibrating capsule on colonic circadian rhythm and bowel symptoms in chronic idiopathic constipation. Neurogastroenterol Motil. 2020 Nov;32(11):e13890. doi: 10.1111/nmo.13890. Epub 2020 May 25. PMID 32449277
- [Background] Ron Y, Halpern Z, Safadi R, Dickman R, Dekel R, Sperber AD. Safety and efficacy of the vibrating capsule, an innovative non-pharmacological treatment modality for chronic constipation. Neurogastroenterol Motil. 2015 Jan;27(1):99-104. doi: 10.1111/nmo.12485. Epub 2014 Dec 6. PMID 25484196
- [Background] Qi Z, Middleton JW, Malcolm A. Bowel Dysfunction in Spinal Cord Injury. Curr Gastroenterol Rep. 2018 Aug 29;20(10):47. doi: 10.1007/s11894-018-0655-4. PMID 30159690